CLINICAL TRIAL: NCT02440919
Title: Effects of Low Oxygen Supplementation and Ventilator Hyperinflation in the Endotracheal Suction of Mechanically Ventilated Patients
Brief Title: Oxygen Supplementation and Ventilator Hyperinflation in the Endotracheal Suction (OSVHES)
Acronym: OSVHES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Jacqueline R F Vianna, Master's degree, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11354813.1.0000.5504
Record Dates: First submitted 2015-03-03; First posted 2015-05-12 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Hypoventilation; Hypoxemia
Keywords: Respiratory mechanics; Oxygenation; Suction; Mechanical ventilation; Respiratory therapy; Capnography; Pulmonary Ventilation
MeSH Terms: conditions — Hypoventilation; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hyperoxygenation - 100% FiO2 (Other): Hyperoxygenation involved supplying 100% fraction of inspired oxygen (FIO2).
  Interventions: Other: Hyperoxygenation 20% FiO2
- Hyperoxygenation - 20% FiO2 (Other): Hyperoxygenation involved supplying 20% oxygen above FiO2 basal.
  Interventions: Other: Hyperoxygenation 100% FiO2
- Hyperinflation - Basal FiO2 (Other): Ventilator hyperinflation, with keeping the oxygen already offered to the patient.
  Interventions: Other: Hyperinflation (PEEP- ZEEP) 20% FiO2
- Hyperinflation - 20% FiO2 (Other): Ventilator hyperinflation and hyperoxygenation involved supplying 20% oxygen.
  Interventions: Other: Hyperoxygenation 20% FiO2; Other: Hyperinflation (PEEP- ZEEP) Basal FiO2

INTERVENTIONS:
Other: Hyperoxygenation 100% FiO2 — Endotracheal suction associated with Hyperoxygenation involved supplying 100% oxygen.
  Arms: Hyperoxygenation - 20% FiO2
Other: Hyperoxygenation 20% FiO2 — Endotracheal suction associated with Hyperoxygenation involved supplying 20% oxygen above FiO2 basal.
  Arms: Hyperinflation - 20% FiO2; Hyperoxygenation - 100% FiO2
Other: Hyperinflation (PEEP- ZEEP) Basal FiO2 — Endotracheal suction associated ventilator hyperinflation (PEEP-ZEEP maneuver) and involved no hyperoxygenation, keeping the oxygen already offered to the patient.
  Arms: Hyperinflation - 20% FiO2
Other: Hyperinflation (PEEP- ZEEP) 20% FiO2 — Endotracheal suction associated ventilator hyperinflation (PEEP-ZEEP maneuver) and hyperoxygenation involved supplying 20% oxygen.
  Arms: Hyperinflation - Basal FiO2

SUMMARY:
This is a double crossover study where all patients are randomly allocated to one of two treatment sequences associated with endotracheal aspiration.The first treatment (A) uses two suctioning methods for each patient: one involving hyperoxygenation with administration of 100% oxygen 1 minute before and after suction (intervention I), and the other hyperoxygenation with oxygen supply to 20% above basal offer (Intervention II) in the same way.The second treatment (B) uses a technique of hyperinflation with the mechanical ventilator (PEEP-ZEEP) associated with hyperoxygenation. The intervention I, uses PEEP-ZEEP offering 20% above basal oxygenation and intervention II uses the PEEP-ZEEP with basal oxygen supply in the same way.

All subjects were randomly allocated using sealed envelopes to a treatment sequence A or B on Day 1. Patients received two treatments, at least four hours apart. The first treatment is in the morning and the alternate treatment is performed in the afternoon. On Day 2 the order of the treatments was reversed using the same patient position sequence.The interventions I and II are performed at least 4 hours apart to minimize any carryover effect.

DETAILED DESCRIPTION:
Endotracheal suction must be carried out only through precise indication, because it is associated with undesirable effects on the hemodynamic parameters, ventilation, oxygenation and respiratory mechanics.

The hyperoxygenation is one of the methods of prevention of hypoxemia induced by tracheal suction procedure and have been proposed for its efficiency. Another method is the hyperinflation with the mechanical ventilator. Ventilator hyperinflation improves oxygenation, mobilizes the bronchial secretion excess and re-expand the lung collapsed areas.

The PEEP-ZEEP is a ventilator hyperinflation technique, described as a lung inflation through a positive pressure enhancement at the end of expiration (PEEP), followed by rapid lung deflation with an abrupt reduction in the PEEP to ZEEP (0 centimeters of water (cmH2O)).

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for more than 12h
* Hemodynamic stability
* Presence of indication criteria of endotracheal aspiration procedure

Exclusion Criteria:

* High doses of vasopressor amines amines and/or severe arrhythmias
* Hemoglobin < 7 g/dL
* FiO2 ≥ 0.6
* PEEP ≥ 10 cmH2O
* Conditions: rib fractures, chest drain, severe bronchospasm, pneumothorax not drained and tracheostomy
* Contraindications of ventilator hyperinflation(PEEP-ZEEP): intracranial pressure > 10 mmHg, bleeding disorders, accented degrees of gastroesophageal reflux and bullous lung disease.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen (SpO2) and Ventilation (ETCO2) measures | Endotracheal suctioning is carried out according each protocol. Oxygen (SpO2) and ventilation (ETCO2) measures are performed before and after supply oxygen given for 1 minute, 60 seconds after each suctioning, immediately after and 30 minutes the end.
  Oxygenation is evaluated by peripheral oxygen saturation (SpO2), measured by a respiratory monitor (DX-2021™ or DX-2023™- Dixtal™. The Impact on oxygenation was detecting hypoxemia with SpO2 values below 90%. Ventilation is evaluated by end-tidal carbon dioxide measured by carbon dioxide sensor (CAPNOSTAT CO2 Sensor, Novametrix Medical Systems Inc.) inserted into the mechanical ventilator circuit Dixtal 3012™ - Dixtal™. The impact on ventilation was detecting hypoventilation with values exceeding 50 mmHg.

SECONDARY OUTCOMES:
Respiratory mechanic measures | Endotracheal suctioning is carried out according each protocol. Baseline Respiratory mechanic measures are performed before suctioning, immediately after and 30 minutes the end.
  Respiratory mechanics was measured by mechanical ventilator Dixtal 3012™- Dixtal™. Its impact will be evaluated by the changes of parameters of normality of variables: auto-PEEP, dynamics compliance (Cd), static compliance (Cst), airway resistance (rva), Airway occlusion pressure (P0.1), slow vital capacity (SVC) and maximal inspiratory pressure (MIP).
Volumetric capnography measures | Endotracheal suctioning is carried out according each protocol. Baseline Volumetric capnography measures are performed before suctioning, immediately after and 30 minutes the end.
  Volumetric capnography was evaluated by carbon dioxide sensor (CAPNOSTAT CO2™ Sensor, Novametrix Medical Systems Inc.) measured by mechanical ventilator Dixtal 3012™- Dixtal™. Its impact will be evaluated by the changes of parameters of normality of variables: ETCO2, anatomical dead space/tidal volume ratio (Vd/VT), alveolar dead space (Vd), alveolar ventilation (Va), maximal tidal elimination of carbon dioxide (VtCO2), carbon dioxide production (VCO2) and partial pressure of expired (PeCO2).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline RF Vianna, Master, Principal Investigator — UFSCar
Locations (1):
- The ICU of Hospital Santa Casa de Misericordia of Batatais, Batatais, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogge JA, Bunde L, Baun MM. Effectiveness of oxygen concentrations of less than 100% before and after endotracheal suction in patients with chronic obstructive pulmonary disease. Heart Lung. 1989 Jan;18(1):64-71. PMID 2912927
- [Background] Berney S, Denehy L. A comparison of the effects of manual and ventilator hyperinflation on static lung compliance and sputum production in intubated and ventilated intensive care patients. Physiother Res Int. 2002;7(2):100-8. doi: 10.1002/pri.246. PMID 12109234
- [Background] Herbst-Rodrigues MV, Carvalho VO, Auler JO Jr, Feltrim MI. PEEP-ZEEP technique: cardiorespiratory repercussions in mechanically ventilated patients submitted to a coronary artery bypass graft surgery. J Cardiothorac Surg. 2011 Sep 13;6:108. doi: 10.1186/1749-8090-6-108. PMID 21914178
- [Derived] de Freitas Vianna JR, Pires Di Lorenzo VA, Lourenco da S Simoes MM, Guerra JL, Jamami M. Effects of Zero PEEP and < 1.0 FIO2 on SpO2 and PETCO2 During Open Endotracheal Suctioning. Respir Care. 2020 Dec;65(12):1805-1814. doi: 10.4187/respcare.07435. Epub 2020 Jul 7. PMID 32636279
- [Derived] Vianna JR, Pires Di Lorenzo VA, Simoes MM, Jamami M. Comparing the Effects of Two Different Levels of Hyperoxygenation on Gas Exchange During Open Endotracheal Suctioning: A Randomized Crossover Study. Respir Care. 2017 Jan;62(1):92-101. doi: 10.4187/respcare.04665. Epub 2016 Nov 15. PMID 28003557